CLINICAL TRIAL: NCT05047744
Title: Dual Mobility Total Joint Prosthesis (Touch) for Thumb Carpometacarpal Joint Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUK-UNF-21-001
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Rhizarthrosis
Keywords: CMC I Osteoarthritis, Total Joint Replacement, Hand Surgery

STUDY DESIGN:
Intervention Model Description: Prospective non randomized Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prosthesis Cohort (Experimental): Surgery dual mobility Prosthesis
  Interventions: Device: Touch Dual Mobility CMC I Prosthesis

INTERVENTIONS:
Device: Touch Dual Mobility CMC I Prosthesis — Surgery

SUMMARY:
The dual mobility concept currently represents the newest generation of thumb carpometacarpal prostheses. The aim of this study was to evaluate the outcomes of TOUCH® prosthesis. From September 2019 to December 2023,a minimum of 100 prosthesis shall be implanted in patients suffering from symptomatic stage III osteoarthritis. All included patients will follow a systematic follow-up regimen (4, 8, 16 weeks, 6, and 12 months as well as 24 months postoperatively).

Radiographics, ROM, VAS, DASH and Pinch grip are measured. Aim of the study is to compare clinical outcome of dual mobility prosthesis with common results of CMC I Prosthesis in literature.

DETAILED DESCRIPTION:
The dual mobility concept currently represents the newest generation of thumb carpometacarpal prostheses. The aim of this study was to evaluate the outcomes of TOUCH® prosthesis. From September 2019 to December 2023,a minimum of 100 prosthesis shall be implanted in patients suffering from symptomatic stage III osteoarthritis. All included patients will follow a systematic follow-up regimen (4, 8, 16 weeks, 6, and 12 months as well as 24 months postoperatively).

Radiographics, ROM, VAS, DASH and Pinch grip are measured. Aim of the study is to compare clinical outcome of dual mobility prosthesis with common results of CMC I Prosthesis in literature.

The Study is designed to give clinical results after one year, 2 years and also long time results in the future.

ELIGIBILITY:
Inclusion Criteria:

* CMC I Osteoarthritis /Stage III)

Exclusion Criteria:

* CMC I (osteoarthritis / Other Stage than III)
* Anticoagulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
DASH Score (Disability of Arm Shoulder and Hand Score) | 24 months
  DASH Score is taken before Surgery and after 6, 12 and 24 months DASH (Disabilty of Arm Shoulder and Hand) Score reaches from 0-100, whereas 0 reprensents best score while 100 represents worst

SECONDARY OUTCOMES:
Subjective Pain | 24 months
  patients report about subjective Pain level in average at 6, 12 and 24 months in a VAS (Visual Analog Pain Scale) scale (0-10), whereas 0 is best and 10 worst

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler Universitaetsklinikum GmbH, Linz, Austria

IPD SHARING:
Plan to Share IPD: Undecided